CLINICAL TRIAL: NCT00780143
Title: Phase I/II Study of Plitidepsin (Aplidin®) in Combination With Cytarabine in Patients With Relapsed/Refractory Leukemia
Brief Title: Clinical Study of Plitidepsin (Aplidin®) in Combination With Cytarabine in Patients With Relapsed/Refractory Leukemia
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: PharmaMar (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APL-A-007-06
Record Dates: First submitted 2008-10-24; First posted 2008-10-27 (Estimated); Results first posted 2018-11-09 (Actual); Last update posted 2018-11-09 (Actual); Status verified 2013-11

CONDITIONS: Relapsed/Refractory Leukemia
Keywords: Tumor; Leukemia; Plitidepsin; Aplidin
MeSH Terms: conditions — Leukemia; Neoplasms | interventions — plitidepsin; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): Plitidepsin in combination with Cytarabine
  Interventions: Drug: Plitidepsin plus Cytarabine

INTERVENTIONS:
Drug: Plitidepsin plus Cytarabine — Plitidepsin 0.54 mg /m2 (initial dose)daily x 5 one hour infusion every 3 weeks plus Cytarabine 1 g/m2 daily for 5 days.

SUMMARY:
This is a Phase I/II study to determine the safety, tolerability and to identify the MTD and DLT of Plitidepsin in combination with a fixed dose of Cytarabine in patients with relapsed/refractory leukemia and to determine the response rate of the combination of Plitidepsin with Cytarabine in patients with relapsed/refractory AML treated at the MTD.

DETAILED DESCRIPTION:
This is a Phase I/II study to determine:

* the safety, tolerability and to identify the MTD and DLT of Plitidepsin in combination with a fixed dose of Cytarabine in patients with relapsed/refractory leukemia and to determine the response rate of the combination of Plitidepsin with Cytarabine in patients with relapsed/refractory AML treated at the MTD.
* the pharmacokinetic parameters of Plitidepsin in combination with Cytarabine.
* whether Plitidepsin in combination with Cytarabine exerts antiangiogenic effects as measured by reduction in microvessel density and VEGFR-1 expression in bone marrow biopsies of patients with relapsed/refractory leukemia.
* whether measurement of free serum VEGF levels, soluble circulating VEGF Receptor and Peripheral Progenitor Endothelial cells provide an early marker of response to Plitidepsin.
* the effects of Plitidepsin and Cytarabine on cytidine deaminase activity and correlate results with Cytarabine drug resistance.
* changes in leukemic gene expression as a result of Plitidepsin and Cytarabine administration.
* tumor response duration.
* progression free survival and overall survival.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have cytologically (or by flow cytometry) documented relapsed/refractory Acute Myeloid leukemia or Acute Lymphoid leukemia for which no standard therapy is anticipated to result in a durable remission. Chronic Myeloid leukemia in blast crisis who progress through Gleevec® or is intolerant to Gleevec® or other FDA approved BCR-ABL Tyrosine Kinase Inhibitors. Patients with untreated AML or ALL who are electing not to receive standard therapy are also eligible. Relapsed/refractory leukemia patients may combination after 1 course of chemotherapy. In addition,leukemia secondary to pre-existing hematologic disorders high-grade myelodysplastic syndromes are also eligible.
2. ≥18 years of age.
3. Patients must be informed of the investigational nature of this study and must give written informed consent in accordance with institutional and federal guidelines.

   Patients who cannot provide informed consent will not be eligible for the study.
4. Prior radiotherapy, chemotherapy or biologic therapies are allowed. Previous line(s) of systemic chemotherapy should have been completed at least 2 weeks prior to starting protocol treatment. Concurrent hydroxyurea administration will be allowed to control WBC count, platelet count, or symptoms and will be discontinued 24 hours prior to the first APLIDIN® dose. For patients with CML in blast crisis, Gleevec® or other BCR-ABL Tyrosine Kinase Inhibitors must be stopped at least 7 days prior to the first APLIDIN® dose. t.
5. Patients must have an ECOG performance status ≤2 (Appendix C).
6. Laboratory data:

   * Serum Total Bilirubin < 1.5 mg/dL X institutional ULN (except when Gilbert syndrome is clearly documented and other LFTs are normal).
   * AST (SGOT)/ALT (SGPT)/ALKP ≤ 2.5 X institutional ULN.
   * Creatinine clearance > 40 ml/min, calculated according to Cockcroft and Gault's formula (Appendix D).
7. Negative pregnancy test for women of childbearing potential.
8. Bone Marrow Assessment within two weeks before the first Aplidin® administration.
9. Estimated life expectancy of > 1 month.
10. Left ventricular ejection fraction within normal limits.

Exclusion Criteria:

1. Previous treatment with Plitidepsin.
2. Prior autologous and/or allogeneic hematopoietic stem cell transplantation (HSCT) patients are not eligible due to higher risk of toxicity related to treatment after such procedure.
3. Active or metastatic secondary primary malignancy.
4. Patients with known Central Nervous System involvement will be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
5. Serious concomitant systemic disorders that would compromise the safety of the patient or compromise the patient's ability to complete the study, including the following specific conditions:

   * Uncontrolled psychiatric illness or medical illness that the principle investigator feels will compromise the patient's tolerance of the study medication.
   * Significant non-neoplastic liver disease (e.g., cirrhosis, active chronic hepatitis).
   * Uncontrolled endocrine diseases (e.g. diabetes mellitus, hypothyroidism or hyperthyroidism) (i.e. requiring relevant changes in medication within the last month, or hospital admission within the last 3 months).
   * Uncontrolled systemic infection.
6. Other relevant cardiac conditions:

   * History or presence of unstable angina, myocardial infarction, valvular heart disease or congestive heart failure.
   * Previous mediastinal radiotherapy.
   * Uncontrolled arterial hypertension despite optimal medical therapy.
   * Previous treatment with doxorubicin at cumulative doses in excess of 400 mg/m².
   * Any grade of cardiac arrhythmia according to CTCAE v3.0 (see appendix F) with exception of < grade 3 supraventricular tachycardia proven to be in response to medical conditions as anemia, fever, etc. from his/her underlying leukemia.
7. History of hypersensitivity reaction to cremophor, Cytarabine, Mannitol, or Plitidepsin (Aplidin®).
8. Myopathy or any clinical situation that causes significant and persistent elevation of CK (> 2.5 ULN in two different determinations performed with one week apart).
9. History of significant Cytarabine related neurotoxicity.
10. Grade >2 motor or sensory neuropathy of any cause.
11. Men and women of reproductive potential who are not using effective contraceptive methods. The effects of Plitidepsin on the developing human fetus at the recommended therapeutic dose are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation and for 6 months after. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. Also, if the wife or female partner of a male patient becomes pregnant during the study, the investigator must be notified promptly and the pregnant woman will be referred for appropriate follow-up with a High-risk Obstetrician.
12. Pregnant and/or lactating women.
13. Patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy, therefore, known HIV-positive patients with active HIV infection and/or receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with Plitidepsin or other agents administered during the study. HIV testing is not required unless infection is clinically suspected.
14. Known active HBV or HCV infection. Patients with any serological evidence of current or past hepatitis B exposure are excluded unless the serological findings are clearly due to vaccination. HBV or HCV testing are not required unless infection is clinically suspected.
15. Concomitant therapy with therapeutic dose of coumadin is not permitted. A suboptimal dose for permeability venous access devices is allowed.
16. Treatment with any investigational product in the 30 days period before inclusion in the study. Wash-out periods since the end of the precedent therapy less than:

    * 6 weeks for nitrosoureas or high dose chemotherapy.
    * 2 weeks for other chemotherapies or biological agents.
    * 4 weeks for radiation or radionuclide therapy (6 weeks in case of prior extensive external beam radiation, more than 25% of bone marrow distribution).
    * 24 hours for hydroxyurea.
    * 7 days for Gleevec® or other BCL-ABL tyrosine Kinase inhibitors.
17. Limitation of the patient´s ability to comply with the treatment or follow-up protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2007-11; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mecide Gharibo, M.D., Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- The Cancer Institute of New Jersey, New Brunswick, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Aplidin®: Plitidepsin in combination with Cytarabine in Patients With Relapsed/Refractory Leukemia
  Plitidepsin plus Cytarabine: Plitidepsin 0.54 mg /m2 (initial dose)daily x 5 one hour infusion every 3 weeks plus Cytarabine 1 g/m2 daily for 5 days.
Period: Overall Study
Arm/Group | Aplidin®
Started | 3
Completed | 0
Not Completed | 3
Not completed — Progressive disease | 1
Not completed — Toxicity | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Aplidin®
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Máximum Tolerate Dose
Description: To determine the maximum tolerated dose (MTD) of Plitidepsin (Aplidin®) when administered daily x 5 days with a fixed dose of Cytarabine for 5 days every four weeks in patients with relapsed/refractory leukemia.
Time Frame: Until disease progression or unacceptable toxicity
Population: The Máximum Tolerate Dose level was not reached
Arm/Group | Aplidin®
Number analyzed (Participants) | 0

2. Primary Outcome: Dose Limiting Toxicity
Description: To determine the dose limiting toxicity (DLT) of Plitidepsin (Aplidin®) when administered daily x 5 days with a fixed dose of Cytarabine for 5 days every four weeks in patients with relapsed/refractory leukemia.
Time Frame: Until disease progression or unacceptable toxicity
Population: The Dose Limiting Toxicity not occurred
Measure: Count of Participants; unit: Participants
Arm/Group | Aplidin®
Number analyzed (Participants) | 3
Participants | 0

3. Primary Outcome: Response Rate
Description: To determine the response rate of the combination of Plitidepsin with Cytarabine in patients with relapsed/refractory AML treated at the MTD.
Time Frame: Until disease progression or unacceptable toxicity
Population: not enough efficacy data were retrieved
Arm/Group | Aplidin®
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Groups:
- Aplidin®: Plitidepsin in combination with Cytarabine
  Plitidepsin plus Cytarabine: Plitidepsin 0.54 mg /m2 (initial dose)daily x 5 one hour infusion every 3 weeks plus Cytarabine 1 g/m2 daily for 5 days.
Arm/Group | Aplidin®
All-Cause Mortality (participants affected / at risk) | 1/3
Serious Adverse Events (participants affected / at risk) | 2/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aplidin® (N=3)
Neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Tachycardia (Cardiac disorders) | 1
Pyrexia (General disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Sepsis (Infections and infestations) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aplidin® (N=3)
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Gingival pain (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Oedema (General disorders) | 1
Tenderness (General disorders) | 1
Sinusitis (Infections and infestations) | 1
Blood alkaline phosphatase increased (Investigations) | 1
Weight decreased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Nocturia (Renal and urinary disorders) | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1
Venous stasis (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days